CLINICAL TRIAL: NCT05574296
Title: Hydrogen's Feasibility and Safety as a Therapy in Extracorporeal Cardiopulmonary Resuscitation
Brief Title: Hydrogen's Feasibility and Safety as a Therapy in ECPR
Acronym: HydrogenFAST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John Kheir, Associate Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-P00043374
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest; Extracorporeal Membrane Oxygenation; Reperfusion Injury
MeSH Terms: conditions — Heart Arrest; Reperfusion Injury | interventions — Hydrogen; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized to usual care with or without treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care + H2 therapy (Experimental): Hydrogen administered via mechanical ventilator and sweep gas into ECMO membrane for 72 hours
  Interventions: Drug: Hydrogen; Other: Usual care
- Usual care (Active Comparator): The current standard of care.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Hydrogen — Hydrogen gas (2%) in air or oxygen administered for 72 hours via ventilator and ECMO membrane. Oxygen concentration titrated per clinical team.
  Other Names: H2 gas
  Arms: Usual care + H2 therapy
Other: Usual care — Usual care post-ECPR event, including targeted temperature management.
  Other Names: Standard of care

SUMMARY:
The purpose of this project is to test the feasibility and safety of inhaled hydrogen gas (H2) administration as a rescue therapy during cardiac arrest requiring extracorporeal cardiopulmonary resuscitation (ECPR, i.e. mechanical circulatory support). Under exemption from informed consent, patients undergoing refractory cardiac arrest in the cardiac ICU at a participating center will be randomized to standard therapy with or without the administration of 2% hydrogen in gases administered via the ventilator and ECMO membrane for 72 hours.

DETAILED DESCRIPTION:
The purpose of this project is to test the feasibility and safety of inhaled hydrogen gas (H2) administration as a rescue therapy during cardiac arrest requiring extracorporeal cardiopulmonary resuscitation (ECPR, i.e. mechanical circulatory support). Each year, 500,000 patients in the US suffer a cardiac arrest and a growing number of them are resuscitated using ECPR. However, neurologic and renal injury remain important resulting comorbidities. The pathophysiology of these often-devastating injuries is ischemia (inadequacy of blood flow, at times compounded by hypoxemia) followed by an abrupt reperfusion (ECMO flow initiation). Among patients with congenital heart disease (CHD) receiving ECPR, 52% either die prior to discharge or suffer severe neurologic impairment. Diatomic hydrogen (H2) administration during and following ECPR may chemically reduce the toxic mediators that directly damage cellular structures and improve neurologically intact survival.

Preclinical data. Several groups have described that H2 inhalation decreases injury when administered following ischemic stroke, myocardial infarction, and cardiac arrest in rodents. Our group demonstrated that inhalation of 2.4% H2 for 24 hours following an experimental swine ischemia-reperfusion injury (as occurs in ECPR) improved neurologic scores, decreased seizures, diminished T2 white matter injury volume by 65%, and improved serum creatinine. Safety study in healthy participants. Under an investigator-initiated IND, we exposed 8 healthy adult participants to up to 72 hours of 2.4% H2 inhalation via high flow nasal cannula, finding no adverse effects on markers of hepatic, renal, cardiac or pulmonary function and no clinically significant symptoms reported. Having received a favorable pre-IND review from the FDA, we propose a two-center early phase study of H2 administration in patients with CHD receiving ECPR.

Study overview. We propose an early-phase randomized trial entitled the 'Hydrogen FAST Trial' (Hydrogen's Feasibility And Safety as a Therapeutic agent). The trial will have a 3-patient vanguard phase and 53 patients with CHD experiencing ECPR randomly assigned in a 3:2 (32/21) ratio to either usual care plus 2% H2 gas for 72 hours or to usual care. Patients will be recruited from two sites. We will primarily examine feasibility and safety (severe adverse events, independently adjudicated), as well as some indicators of efficacy.

Hypotheses. Primary feasibility endpoint: We hypothesize that H2 gas will be administered for a mean of >90% of the first 72 consecutive post-arrest hours in patients so-assigned. Primary safety endpoint: We hypothesize that compared with patients receiving usual post-arrest care, patients receiving H2 will not exceed the treatment-related SAE rate of the usual care group by >12.5% in the 30 days following randomization. Secondary feasibility endpoint: We hypothesize that H2 gas will be administered for a mean of >90% of the first 72 consecutive hours post-H2 initiation in patients so-assigned.

ELIGIBILITY:
INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Patients admitted to a cardiac intensive care unit at a participating site with cardiac comorbidity, including congenital heart disease, myocarditis, cardiac arrhythmia, or rejection of a transplanted heart.
2. Patients are anticipated to be between birth to 18 years of age, although occasionally a patient over the age of 18 may be enrolled.
3. Patient experiencing a refractory cardiac arrest >5 minutes and receiving ongoing CPR in the ICU, cardiac catheterization lab, or cardiac operating room.
4. The decision made by the clinical team to resuscitate from ongoing, refractory cardiac arrest using ECPR due to a lack of other available options.

EXCLUSION CRITERIA

Meeting any of the following criterion renders the patient ineligible for the trial:

1. Enrollment in the opt-out program.
2. Patients known to be pregnant.
3. Patients who are prisoners.
4. Prior ECPR episode during admission (whether or not they were enrolled in the trial).
5. Enrollment does not occur within 6 hours of the decision to resuscitate using ECPR.

Note that ECMO cannulation without preceding CPR does not qualify as ECPR and such patients will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of hydrogen administration (primary) | 72 hours
  Percentage of the first 72 consecutive post-arrest hours (starting at the time of first CPR initiation) in which H2 gas was administered via all of the applicable pathways (e.g. mechanical ventilator and ECMO membrane).
Safety of hydrogen administration | 30 days
  Incidence rate of SAEs of interest per day during the first 30 days post-randomization that have been classified as treatment-related or possibly treatment-related.

SECONDARY OUTCOMES:
Survival to hospital discharge | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Survival to hospital discharge
ICU length of stay | From date of randomization until the date of first ICU discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Duration of ICU stay until first transfer out of ICU
Hospital length of stay | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Duration of hospital stay until first hospital discharge
Functional status score | Calculated on admission to the hospital, at 24 h before cardiac arrest, at hospital discharge, and at 6 months post-randomization
  Functional status score computed based on a detailed review of neurology notes, primary team notes, nursing notes and physical exam documentation by two independent investigators.
Feasibility of hydrogen administration (secondary) | 72 hours
  Percentage of the first 72 consecutive hours post-H2 initiation in which H2 gas was administered via all of the applicable pathways (e.g. mechanical ventilator and ECMO membrane).

CONTACTS AND LOCATIONS:
Overall Officials: John N Kheir, MD, Principal Investigator — Associate Professor of Pediatrics, Harvard Medical School
Locations (4):
- United States (4):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habet V, DeWaard T, Boggs KM, Fetch A, Puente BN, Sleeper LA, Kheir JN. Hydrogen's Feasibility and Safety as a Therapy in Extracorporeal Cardiopulmonary Resuscitation (Hydrogen-FAST): study protocol for a trial of inhaled hydrogen gas as an adjunctive therapy in refractory cardiac arrest. Trials. 2025 Nov 7;26(1):481. doi: 10.1186/s13063-025-09217-7. PMID 41204320